CLINICAL TRIAL: NCT01220700
Title: Antimicrobial Coated Sutures in Paediatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oulu (Other)
Responsible Party: Principal Investigator, Marjo Renko, docent, University of Oulu
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Triclosan
Record Dates: First submitted 2010-10-12; First posted 2010-10-14 (Estimated); Last update posted 2015-02-06 (Estimated); Status verified 2015-02

CONDITIONS: Wound Infections
MeSH Terms: conditions — Wound Infection | interventions — Polyglactin 910

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Triclosane (Experimental): triclosan coated suture material
  Interventions: Other: Triclosane
- Control (Active Comparator): ordinary suture material
  Interventions: Other: Control

INTERVENTIONS:
Other: Triclosane — Triclosane coated suture material
  Other Names: Vicryl plus
  Arms: Triclosane
Other: Control — Ordinary suture material
  Other Names: Vicryl
  Arms: Control

SUMMARY:
The purpose of this study is to determine if suture material coated by antimicrobial agent triclosan would decrease the incidence of surgical site infections (SSIs) in paediatric surgery compared to ordinary sutures.

1500 children (age form 4 weeks to 18 years) coming for general pediatric surgery to the Oulu University Hospital are randomised to have sutures coated with triclosan (Vicryl Plus, Monocryl Plus) or ordinary sutures. The occurrence of SSIs is monitored by email questionnaires to the parents on days 10 and 30. The diagnosis of SSIs are made along CDC criteria.

DETAILED DESCRIPTION:
We have now (spring 2014) recruited almost 1500 patients to the study. When reviewing the recruited material, we found out that the study suture material has been used in 83% of the recruited patients. The reasons for this have been clinical issue during the operation where melting suture material may not have been needed at all.

We have decided to prolong recruiting so that we would gather the calculated sample size of 1500 of patient with study suture material. This will take 12-18 months (probably till autumn 2015).

ELIGIBILITY:
Inclusion Criteria:

* any general surgery during childhood where melting sutures will be used

Exclusion Criteria:

* wound infection as a cause for surgery

Ages: 4 Weeks to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1635 (Actual)
Dates: Start 2010-09; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
occurrence of surgical site infections | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Marjo Renko, MD, PhD, Principal Investigator — University of Oulu, Department of Paediatrics; Terhi Tapiainen, MD, PhD, Study Chair — University of Oulu, Deparment of Paediatrics; Willy Serlo, prof, Study Chair — University of Oulu, Deparment of Peadiatric Surgery; Matti Uhari, prof, Study Director — University of Oulu, Department of Paediatrics; Juha-Jaakko Sinikumpu, MD, Study Chair — University of Oulu, Department of Paediatric Surgery
Locations (1):
- Oulu University Hospital/ Paediatric Surgery, Oulu, Finland

REFERENCES:
- [Derived] Renko M, Paalanne N, Tapiainen T, Hinkkainen M, Pokka T, Kinnula S, Sinikumpu JJ, Uhari M, Serlo W. Triclosan-containing sutures versus ordinary sutures for reducing surgical site infections in children: a double-blind, randomised controlled trial. Lancet Infect Dis. 2017 Jan;17(1):50-57. doi: 10.1016/S1473-3099(16)30373-5. Epub 2016 Sep 19. PMID 27658562